CLINICAL TRIAL: NCT05422573
Title: Randomized Clinical Trial of the Sequence of Genetic Counseling and Testing to Optimize Efficiency, Patient Empowerment and Engagement, and Medical Adherence for Diverse Genetic Testing Indications
Brief Title: Clinical Trial of the Sequence of Cardiovascular Genetic Counseling and Testing
Acronym: RESEQUENCEGC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00320656; R01HG011902 (NIH)
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Genetic Counseling; Inherited Cardiac Disease
Keywords: inherited heart disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (No Intervention): Pre-test genetic counseling appointment with results returned by phone or EHR. Post-test appointment available upon request.
- Efficiency (Experimental): Pre-test genetics education by educational video with an OPTIONAL call with a genetic counselor to address questions. Pre-test appointment available by request. Post-test genetic counseling appointment.
  Interventions: Behavioral: post-test cardiovascular genetic counseling with pre-test education by video; Behavioral: optional phone call with genetic counselor pre-test
- Flipped (Experimental): Pre-test genetics education by educational video with a REQUIRED call with a genetic counselor to address questions. Pre-test appointment available by request. Post-test genetic counseling appointment.
  Interventions: Behavioral: post-test cardiovascular genetic counseling with pre-test education by video; Behavioral: required phone call with genetic counselor pre-test

INTERVENTIONS:
Behavioral: post-test cardiovascular genetic counseling with pre-test education by video — post-test cardiovascular genetic counseling with pre-test education by video
  Arms: Efficiency; Flipped
Behavioral: required phone call with genetic counselor pre-test — REQUIRED phone call with genetic counselor pre-test.
  Arms: Flipped
Behavioral: optional phone call with genetic counselor pre-test — OPTIONAL phone call with genetic counselor pre-test
  Arms: Efficiency

SUMMARY:
Although pre-test genetic counseling is widely recommended and has come to dominate genetic counseling practice, tailored results-focused genetic counseling could both increase genetic counseling efficiency and improve genetic counseling outcomes for the growing number of patients seeking genetic testing for recommended genome-guided medical management. This study will test that hypothesis in adults referred for cardiovascular genetic counseling and testing at the Johns Hopkins Center for Inherited Heart Diseases. This study is a three-arm randomized clinical trial to evaluate two complementary approaches to shifting the primary genetic counseling session to post-test for 510 adults with two broad cardiovascular genetic counseling indications: diagnostic panel testing and family-specific variant testing. The investigators will compare usual care (pre-test genetic counseling appointment, results returned by phone / electronic health record) with online video-based pre-test tailored genetic education with an optional (efficiency arm) or required (flipped arm) phone call with a genetic counselor followed by a post-test genetic counseling appointment. The investigators hypothesize that post-test genetic counseling will: 1) increase efficiency, 2) promote patient empowerment and adherence, and 3) have similar genetic test-associated psychosocial impact.

DETAILED DESCRIPTION:
This is a three-arm randomized clinical trial with a parallel-group design comparing usual care (pre-test genetic counseling, test results by phone/electronic health record (EHR)) to two approaches to post-test results-focused genetic counseling involving a pre-test educational video with an optional [efficiency arm] or required [flipped arm] phone call with a genetic counselor followed by a post-test genetic counseling appointment. Consented participants will be randomly allocated to the three study arms stratified by genetic testing indication (cardiovascular panel, family-specific variant). Questionnaires will be administered at 4 timepoints: 2 weeks before pre-test education/counseling (Q1), immediately after pre-test education/counseling and test ordered or declined (Q2), 2-weeks post-disclosure (Q3), and 6-months post-disclosure (Q4) (Aims 1-3). Data will be extracted from each participant's electronic health record (EHR) to record potential clinical covariates (Aims 1-3), validate self-reported adherence to medical recommendations (Aim 3), and obtain metrics to measure genetic counseling efficiency (Aim 4).

ELIGIBILITY:
Inclusion Criteria:

Cardiovascular panel testing inclusion criteria:

1. Adult (age 18+) scheduled for outpatient genetic counseling in the Johns Hopkins Center for Inherited Heart Diseases,
2. Clinical diagnosis or suspected clinical diagnosis of a potentially inherited cardiovascular disease including a) hypertrophic, dilated, or arrhythmogenic cardiomyopathy, b) ventricular or atrial arrhythmias or an ECG-pattern suspicious for an inherited cardiovascular disease including catecholaminergic polymorphic ventricular tachycardia, long QT syndrome, or Brugada syndrome, or c) a diagnosed or suspected lipid disorder or early-onset coronary artery disease,
3. next-generation cardiovascular sequencing panel clinically indicated.

Family specific variant testing inclusion criteria:

1. Adult (age 18+) scheduled for outpatient genetic counseling in the Johns Hopkins Center for Inherited Heart Diseases,
2. Documented pathogenic or likely pathogenic variant in a gene associated with a hereditary cardiomyopathy, arrhythmia syndrome, or lipid disease in a family member,
3. Referred to the Center for Inherited Heart Diseases for family-specific variant testing.

Exclusion Criteria:

1. Previous genetic counseling at Johns Hopkins for this clinical indication,
2. Previous genetic testing that definitively identified the genetic cause of the patient's condition,
3. Patient unable to speak or read English,
4. Genetic counseling appointment is not anticipated to include genetic testing (for instance if it was scheduled to discuss family communication or adaptation to a new diagnosis),
5. Next generation sequencing panel not clinically indicated (panel cohort only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in empowerment as measured on the Genetic Counseling Outcomes Scale (GCOS) | Baseline up to 2-weeks after genetic counseling result appointment / disclosure
  Change in empowerment as measured on the Genetic Counseling Outcomes Scale (GCOS). The GCOS is 24-item Likert scale with a 7-item response set. Scores range from 24-168 with higher scores indicating higher empowerment.
Anxiety as measured on the Hospital Anxiety and Depression Scale (HADS) | 6-months post results disclosure
  Anxiety as measured on the Hospital Anxiety and Depression Scale (HADS). The HADS contains 14 items measured on a 4-point Likert scale. The anxiety subscale contains 7 items. HADS subscale scores ≥8 indicate potentially clinically significant anxiety and depression and scores ≥10 a likely case.
Medical adherence as assessed by proportion of completed screening tests | 6-months post results disclosure
  Proportion of recommended cardiology appointments and screening tests completed or scheduled
Efficiency as assessed by minutes of counseling time | Up to 6-months post results disclosure
  Total minutes of counseling time per patient documented in the electronic health record including visit and phone notes.

SECONDARY OUTCOMES:
Change in engagement as assessed by Patient Activation Measure | Baseline, 6-months post results disclosure
  Change in patient engagement as measured by the short form of the Patient Activation Measure (PAM-13). The PAM-13 includes a 4-item Likert scale response set with higher scores indicating higher patient activation. To calculate the total PAM score, the raw score is divided by the number of items answered (excepting non-applicable items) and multiplied by 13. Then, this score is transformed to a scale with a theoretical range 0-100, based on calibration tables, with higher PAM scores indicating higher patient activation.
Informed Choice as assessed by Multidimensional Model of informed Choice pilot scales | up to 14 days post-education
  Multidimensional Model of informed Choice pilot scales for familial hypercholesterolemia (FH) and cardiomyopathy/arrhythmia testing will be used. This is a scale that combines a subscale with 8 True/false knowledge about cardiovascular genetics and genetic testing questions scored as number correct with a 5-item scale with a Likert scale response set assessing attitudes toward genetic testing. The entire scale is scored by combining knowledge, values and testing choice made.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia James, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No